CLINICAL TRIAL: NCT05196295
Title: To Evaluate the Safety of Treating Rheumatologic and Metabolic Patients With 3 Increasing Doses of Molecular Hydrogen Supplement.
Brief Title: To Evaluate the Safety of Treating Rheumatologic and Metabolic Patients With Molecular Hydrogen Supplement.
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: HoHo Biotech (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2021007-A
Record Dates: First submitted 2022-01-03; First posted 2022-01-19 (Actual); Last update posted 2022-02-10 (Actual); Status verified 2022-01

CONDITIONS: Autoimmune Diseases; Metabolic Disease
MeSH Terms: conditions — Autoimmune Diseases; Metabolic Diseases | interventions — Hydrogen

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Hydrogen capsules (Experimental): Participants will be allocated by doctors and receive either 1 (n=5), 3 (n=5) or 6 (n=5) capsules every day for one month.
  Interventions: Drug: Hydrogen

INTERVENTIONS:
Drug: Hydrogen — Participants take either 1 (n=5), 3 (n=5) or 6 (n=5) capsules every day for one month.

SUMMARY:
The latest international research shows that supplementation of hydrogen molecules as an aid, adjuvant, can speed up the course of the disease. The purpose of this study is to determine the safety and possible efficacy of hydrogen supplements in different dose exposures for a clinical study in rheumatologic and metabolic patients. Patients will receive a different dosage of hydrogen capsules with their conventional treatment for a month. Investigators will test for any changes in haematologic, urine analysis and health status during and following the exposure period.

DETAILED DESCRIPTION:
According to the current literature, there is a lack of specific drugs for chronic inflammatory symptoms which develop from many refractory diseases with complicated clinical features. Hydrogen supplement has been shown to have significant removal effects on free radicals and reduce chronic inflammation. With these benefits, molecular hydrogen may have the ability to speed up the recovering the disease.

The purpose of this study is to determine the safety and possible efficacy of hydrogen supplements in the different doses of hydrogen capsules for a clinical study in rheumatologic and metabolic patients.

Study design: 15 rheumatologic patients and 15 metabolic patients will be recruited from the Min-Sheng General Hospital for this study. Participants will be screened by doctors for their eligibility and undergo a series of tests (questionnaires and examinations). Consenting participants will then be allocated into 3 groups by different dosage (Low, n=5; Medium, n=5; High, n=5). Participants will receive 1 (Low), 3 (Medium) or 6 (High) capsules every day for one month. Participants will be examined their regular haematology, urine and health status before and after the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Age 20 to 70 with autoimmune or metabolic diseases
* Able to compliant with the protocol
* Able to return to the hospital regularly

Exclusion Criteria:

* Pregnancy
* Expected pregnancy

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-01-11 (Actual); Primary Completion 2022-07-30 (Estimated); Study Completion 2022-07-30 (Estimated)

PRIMARY OUTCOMES:
Adverse effects/symptoms | up to 28 days
  Any adverse effects will be codified according the the NCI CTCAE v5.0

SECONDARY OUTCOMES:
Change in physiological parameter (Blood Routine) | Change from Baseline Blood Routine at Day 28
  Numerical change in Blood Routine
Change in physiological parameter (Urine Routine) | Change from Baseline Urine Routine at Day 28
  Numerical change in Urine Routine
Brief Fatigue Inventory-Taiwan (BFI-T) (6 questions) | Change from Baseline BFI-T at Day 28
  Questionnaire for rheumatologic patients minimum values:0 maximum values:60 Higher scores mean a worse outcome.
Control status scale for diabetics (CSSD70) (First part: 11 questions) | Change from Baseline CSSD70 at Day 28
  Questionnaire for metabolic patients minimum values:0 maximum values:22 Higher scores mean a worse outcome.

CONTACTS AND LOCATIONS:
Locations (1):
- Min-Sheng Gereral hospital, Taoyuan District, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Chiu SH, Douglas FL, Chung JR, Wang KY, Chu CF, Chou HY, Huang WC, Wang TY, Chen WW, Shen MC, Liu FC, Hsiao PJ. Evaluation of the safety and potential lipid-lowering effects of oral hydrogen-rich coral calcium (HRCC) capsules in patients with metabolic syndrome: a prospective case series study. Front Nutr. 2023 Jul 14;10:1198524. doi: 10.3389/fnut.2023.1198524. eCollection 2023. PMID 37521410